CLINICAL TRIAL: NCT01526772
Title: A Prospective Study Evaluating The Utility of Transnasal Endoscopy With Roux en Y Gastric Bypass Referred for Upper Endoscopy
Brief Title: A Prospective Study Evaluating The Utility of Transnasal Endoscopy With Roux en Y Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00018487
Record Dates: First submitted 2012-01-17; First posted 2012-02-06 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: Transnasal; Transoral; Roux en Y gastric bypass; Upper Endoscopy; Obesity
MeSH Terms: conditions — Obesity | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who have undergone RYGB: Patients who have undergone RYGB and have been referred for an EGD
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Transoral endoscopy versus transoral endoscopy
  Other Names: Endoscopy performed transnasally with a slim scope; Transoral endoscopy with a routine diagnostic endoscope

SUMMARY:
Improvements in imaging technology have allowed for the development of small endoscopes ("slim scopes") half the size of a typical endoscope. These small endoscopes can be passed transnasally into the esophagus and stomach with only local anesthesia to the nasal passage without the need for deep sedation. They have been used in the detection of diseases of the esophagus and stomach,3,4 but have not been used in the detection of complications in the post bariatric population

DETAILED DESCRIPTION:
Obesity is an epidemic in the United States effecting 250 million people worldwide and over 30% of the population of the United Sates. Medical therapy for obesity is lacking in its durability in maintaining weight loss. Currently surgical therapy is the most dependable and durable treatment option. The Roux en Y gastric bypass (RYGB) was initially described in 1967 and is currently the surgical method of choice in the treatment of obesity. It involves the creation of a small gastric pouch by restricting the gastric body and antrum and the creation of a long roux limb with a gastrojejunal anastomosis, thus inducing satiety and creating a malabsorptive physiology. Unfortunately this procedure maintains a significant complication rate. Strictures at the gastrojejunal anastomosis occur in 6-20% of patients after bypass.1 Anastomotic ulcers occur in up to 16% .2 Symptoms include vomiting, abdominal pain, and significant nausea. Unfortunately these symptoms are not specific to strictures or ulcers and may occur spontaneously without a specific etiology, so often a transoral upper endoscopy (EGD) is required to evaluate the anastomosis for significant pathology.

EGD in post bariatric patients is a safe procedure. However it typically requires deep sedation administered by an anesthesiologist to overcome the patient's gag reflex and discomfort. Sedation in obese patients can be challenging due to the risks of apnea and challenges of tracheal intubation. For the procedure to be performed the patient must take the day off from work and bring a driver to take them home, thus there are significant direct and indirect costs to the procedure.

Improvements in imaging technology have allowed for the development of small endoscopes ("slim scopes") half the size of a typical endoscope. These small endoscopes can be passed transnasally into the esophagus and stomach with only local anesthesia to the nasal passage without the need for deep sedation. They have been used in the detection of diseases of the esophagus and stomach,3,4 but have not been used in the detection of complications in the post bariatric population

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to review and sign informed consent
* Subjects have undergone Roux en Y gastric bypass
* Subjects report any of the following symptoms that would prompt investigation and referral for an upper endoscopy; abdominal pain, nausea, vomiting or problems swallowing

Exclusion Criteria:

* Patients who cannot give and sign informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This pilot study will attempt to recruit 20 subjects over one year.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07-07 (Actual); Study Completion 2014-07-07 (Actual)

PRIMARY OUTCOMES:
Anastomotic ulcer and diameter | 1 year
  Presence of anastomic ulcer seen by slim scope

SECONDARY OUTCOMES:
Presence of anastomotic stricture and diameter | 1 years
  Presence of anastomotic sticture seen by slim scope and estimated anastomis diameter

CONTACTS AND LOCATIONS:
Overall Officials: John O Evans, MD, Principal Investigator — Wake Forest University Baptist Health
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States